CLINICAL TRIAL: NCT00940095
Title: A Prospective, Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Efficacy and Safety of Clazosentan in Reducing Vasospasm-related Morbidity and All-cause Mortality in Adult Patients With Aneurysmal Subarachnoid Hemorrhage Treated by Endovascular Coiling.
Brief Title: Clazosentan in Aneurysmal Subarachnoid Hemorrhage
Acronym: CONSCIOUS-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy data from the Phase 3 clinical study (AC-054-301; CONSCIOUS-2)
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-054-302
Record Dates: First submitted 2009-07-13; First posted 2009-07-15 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: Subarachnoid; Aneurysmal; surgical clipping; PIVLAZ; vasospasm; cerebral vasospasm; clazosentan; Actelion; Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial; Hemorrhage | interventions — clazosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Clazosentan 5 mg/h (Experimental): Continuous intravenous infusion of clazosentan (5 mg/h) started within 56 hours post-aSAH and scheduled to continue until Day 14 post-aSAH, or at least until Day 10 post-aSAH, for patients discharged before Day 14
  Interventions: Drug: Clazosentan 5 m/h
- Clazosentan 15 mg/h (Experimental): Continuous intravenous infusion of clazosentan (15 mg/h) started within 56 hours post-aSAH and scheduled to continue until Day 14 post-aSAH, or at least until Day 10 post-aSAH, for patients discharged before Day 14
  Interventions: Drug: Clazosentan 15 mg/h
- Placebo (Placebo Comparator): Continuous intravenous infusion of placebo matching clazosentan started within 56 hours post-aSAH and scheduled to continue until Day 14 post-aSAH, or at least until Day 10 post-aSAH, for patients discharged before Day 14
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clazosentan 5 m/h — Continuous intravenous infusion of clazosentan (5 mg/h)
  Other Names: ACT-108475 (AXV-034343)
  Arms: Clazosentan 5 mg/h
Drug: Clazosentan 15 mg/h — Continuous intravenous infusion of clazosentan clazosentan (15 mg/h)
  Other Names: ACT-108475 (AXV-034343)
  Arms: Clazosentan 15 mg/h
Drug: Placebo — Continuous intravenous infusion of placebo-matching clazosentan
  Arms: Placebo

SUMMARY:
The aim of this study is to demonstrate that clazosentan, administered as a continuous intravenous infusion at either 5 mg/h or 15 mg/h until Day 14 post aneurysmal subarachnoid hemorrhage (aSAH), reduces the incidence of cerebral vasospasm-related morbidity and all-cause mortality within 6 weeks post-aSAH treated by endovascular coiling.

The primary endpoint of the study is the occurrence of cerebral vasospasm-related morbidity, and mortality of all-causes within 6 weeks post-aSAH, defined by at least one of the following:

1. Death (all causes).
2. New cerebral infarct(s) due to cerebral vasospasm as either the primary or relevant contributing cause, or not adjudicated to be entirely due to causes other than vasospasm.
3. Delayed ischemic neurological deficit (DIND) due to cerebral vasospasm as either the primary or relevant contributing cause, or not adjudicated to be entirely due to causes other than vasospasm.
4. Administration of a valid rescue therapy in the presence of confirmed cerebral vasospasm on angiography (DSA or CTA).

An independent Critical Events Committee (CEC) will adjudicate whether or not patients meet the primary endpoint and its individual morbidity components.

ELIGIBILITY:
Inclusion Criteria :

1. Males and females aged 18 to 75 years (inclusive).
2. Patients with a ruptured saccular aneurysm, confirmed by angiography (digital subtraction angiography [DSA] or computed tomography angiography [CTA], investigator's assessment), and which has been successfully* secured by endovascular coiling. The time of aneurysm rupture must be known or possible to estimate with a reasonable degree of certainty.
3. World Federation of Neurological Surgeons (WFNS) grade I-IV measured prior to the endovascular coiling procedure, and which does not worsen to grade V post-procedure (based on regular Glasgow Coma Scale [GCS])
4. Patients with any thick clot (short axis > or = 4 mm) on baseline CT scan (investigator's assessment).
5. Women of childbearing potential must have a negative serum pregnancy test and must use a reliable method of contraception during the 12 weeks following study drug discontinuation.
6. Written informed consent to participate in the study must be obtained from the patient or a legal representative prior to initiation of any study-mandated procedure and randomization.

Exclusion Criteria :

1. Subarachnoid hemorrhage (SAH) due to causes other than saccular aneurysm.
2. Giant aneurysms (height or width > or = 25 mm).
3. Intraventricular or intracerebral blood, in absence of subarachnoid blood, or or with only a thin clot (short axis < 4 mm)
4. Cerebral vasospasm on angiography (investigator's assessment) prior to endovascular coiling (intraprocedural cerebral vasospasm is not an exclusion criterion).
5. A major complication during the endovascular coiling procedure, such as massive intracranial bleeding, intracranial thromboembolism, coil migration, aneurysm perforation or rupture, arterial dissection, major arterial occlusion, a large territorial cerebral infarct defined as involving > 1/3 of a vascular territory, or a new major neurological deficit post-procedure (e.g., hemiplegia or aphasia lasting > or = 12 hours post-aneurysm coiling)*.
6. Current ruptured aneurysm previously secured (successfully or not) by clipping.
7. Coiling material used, which has not been approved by local health authorities.
8. Use of liquid embolism aneurysmal treatment or flow diverting device.
9. Several aneurysms among which the ruptured one cannot be identified with certainty and which are not all secured during the coiling procedure.
10. No end-of-procedure DSA.
11. Another securing procedure planned for any aneurysm between randomization and Week 12 post-aSAH.
12. Study drug start >56 hours after the aneurysm rupture.
13. Known, at time of screening, that certain follow-up, or protocol-mandated imaging assessments will not be feasible.
14. Hypotension (systolic blood pressure < or = 90 mmHg) refractory to treatment.
15. Aspiration pneumonia.
16. Pulmonary edema or severe cardiac failure requiring inotropic support at time of randomization.
17. Any severe or unstable concomitant condition or disease (e.g., known significant neurological deficit, cancer, hematological, coronary disease, psychiatric disorder), which would affect assessment of the safety or efficacy of the study drug (investigator's opinion).
18. Significant kidney disease defined by plasma creatinine > or = 2.5 mg/dL (221 micromol/l) and/or liver disease defined by total bilirubin > 2-fold Upper Limit of Normal as measured at local laboratory, and/or known diagnosis or clinical suspicion of liver cirrhosis.
19. Infusion of i.v. nimodipine or i.v. nicardipine must have these drugs discontinued at least 4 hours prior to initiation of study treatment.
20. Infusion of i.v. fasudil within 24-hour period preceding planned start of study drug initiation.
21. Start of statins less than 2 weeks prior to admission must have them discontinued prior to study drug initiation.
22. Infusion of cyclosporin A or other calcineurin inhibitors (e.g., tacrolimus), or patients for whom it is known at the time of randomization that these medications will be started during the study drug infusion period.
23. Intake of an investigational product including investigational coil material within 28 days prior to randomization or those who have already participated in current study or CONSCIOUS-2 (AC-054-301).
24. Unlikely event to comply with protocol (e.g., unable to return for follow-up visits).
25. Known hypersensitivity to other endothelin receptor antagonists.26.current alcohol or drug abuse/dependence.

    * "Large territorial infarct" refers to infarcts detected during the endovascular coiling procedure or immediately post-procedure (i.e., CT performed for suspicion of cerebral infarct or other complication). This does not imply having to wait 24-48 hours post-procedure to perform the protocol-mandated CT scan in order to randomize a patient. Evaluation for a new major neurological deficit post-procedure implies reversal of sedation and performance of a GCS examination (verbal scores in intubated patients may be extrapolated from the eye-opening and motor scores using predefined values). If a new major neurological deficit does not improve within 12 hours after the coiling procedure, the patient cannot be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2009-07-01; Primary Completion 2010-10-01 (Actual); Study Completion 2011-01-01 (Actual)

PRIMARY OUTCOMES:
Cerebral vasospasm-related morbidity and mortality of all-causes as defined by the protocol | Within 6 weeks post-aSAH

SECONDARY OUTCOMES:
Glasgow Outcome Scale Extended (GOSE) at Week 12 post-aSAH, dichotomized into good (score > 4) and poor (score ≤ 4) outcome. | Week 12 post-aSAH

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Roux, MD, Study Director — Actelion
Locations (144):
- United States (29):
  - Glendale Adventist Medical Center, Glendale, California
  - UCSF Medical Centre, San Francisco, California
  - Stanford Hospital and Clinis, Stanford, California
  - Colorado Neurological Institute, Englewood, Colorado
  - Yale Univerity School of Medicine, New Haven, Connecticut
  - University of South Florida, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Illnois, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Centre, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Barnes_Jewish Hospital, St Louis, Missouri
  - Capital Health System Inc. d/b/a The Stroke and Cerebrovascular Center of New Jersey, Trenton, New Jersey
  - Columbia University Medical Center, New York, New York
  - New York Presbyteruan Hospital - Weill Cornell Medical Centre, New York, New York
  - State University of New York at Stony Brook, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Thomas Jefferson University School of Medicine, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Zale Lipshy Hospital, Dallas, Texas
  - Univ. of VA Health System, Charlottesville, Virginia
  - Virginia Commonwealth University Medical Centre, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Argentina (3):
  - Hospital Aleman, Buenos Aires
  - Clinica De Sol, Buenos Aires
  - ENERI, Buenos Aires
- Australia (5):
  - Gold Coast Hospital, Southport, Queensland
  - Royal Brisbane & Women's Hosptal, Brisbane
  - Royal Prince Alfred Hosptial, Camperdown
  - Monash Medical Centre, Clayton
  - Princess Alexandra Hospital, Woolloongabba
- Austria (4):
  - Landeskrankenhaus und Medizinische Universitat, Graz
  - Medizinsche Universitat Innsbruck, Innsbruck
  - University Fur Neurochirurgie, SALK, Christian Doppler Hospital, Salzburg
  - AKH University of Vienna, Medical Univ. Of Neurosurgery, Vienna
- Belgium (6):
  - UZ Antwerpen, Antwerp
  - ULB Erasme, Brussels
  - UZ Brussels, Brussels
  - UCL Saint-Luc, Brussels
  - UZ Gent, Ghent
  - UZ Gasthuisberg, Leuven
- Brazil (7):
  - Hospital das Clinicas da UFMG, Belo Horizonte
  - Hospital de Clinicas da Universidade Federal do Parana, Curitiba
  - Clinica de Neurologia de, Joinville
  - Hospital de Clínicas de Niteroí, Niteroí
  - Hospital Moinhos de Vento, Porto Alegre
  - Hospital Santa Marcelina, São Paulo
  - Santa Case de Misericordia de Sobral, Sobral
- Canada (9):
  - University of Calgary - Foothills Medical Center, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver Hospital & Health Sciences, Vancouver, British Columbia
  - QEII Heath Sciences Center - Halifax Infirmary, Halifax, Nova Scotia
  - Hamilton General Hospital, Toronto, Ontario
  - St. Michael's Hospital, University of Toronto, Toronto, Ontario
  - CHUM Hospital - Notre Dame, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Hopital de I'Enfant-Jesus, Québec
- Chile (5):
  - Hospital Regional de Concepción, Concepción
  - Institute de Neurocirugia, Santiago
  - Hospital Clinico Pontificia Universidad Católica de Chile, Santiago
  - Clinica Davila, Santiago
  - Hospital Carlos Van Buren, Valparaíso
- Czechia (8):
  - Fakultni nemocnice Bmo, Brno
  - Nemocnice Ceske Budejovice, České Budějovice
  - Fakultní nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Ostrava, Ostrava
  - Nemocnice Na Homolce, Prague
  - ÚVN Praha, Prague
  - Fakultni nemocnice Homoice, Prague
  - Masarykova nemocnice Usti n. Labem, Ústí nad Labem
- Denmark (3):
  - The Neuroscience Center, Copenhagen University Hospital, Copenhagen
  - Glostrup Hospital, Glostrup Municipality
  - Odense University Hospital, Odense
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Tampere University Central Hospital (TAYS), Tampere
- France (8):
  - CHU d'Angers, Angers
  - Hopital Pellegrin, Bordeaux
  - Hopital neurologique et Neuro-Chirurgical Pierre Wertheimer, Bron
  - Hopital Henru Mondor, Créteil
  - Hopital General, Dijon
  - Hopital de la Timone - CHU de Marseille, Marseille
  - Hopital Gui de Chauliac, Montpellier
  - Hopital central, Nancy
- Germany (14):
  - Universitatsklinikum Augsburg Clinic for Diagnostic Radiology and Neuroradiology, Augsburg
  - Charite Universitatsmedzin Berlin, Berlin
  - Universitatsklinikum Bonn, Bonn
  - University of Bonn Medical Center, Bonn
  - Klinik imd Poliklinik fur Neurochirurgie, Dresden
  - Universitaet Erlangen-Nuerberg Klinik fur Neurologie, Erlangen
  - University Hospital of Essen, Essen
  - Universitatsklinik Frankfurt, Klinik und Poliklinik f. Neurochirurgie, Frankfurt
  - Neuroradiologie der Universitatsklinik Freiburg, Freiburg im Breisgau
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Neurochirurggische Universitatsklinik des Heidelberg, Heidelberg
  - Klinik und Poliklinik fur Neurochirurgie, Leipzig
  - Thechnical University - Klinikum rechts der Isar, Munich
  - University Regensburg, Regensburg
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince od Wales Hospital, Shatin
- Hungary (3):
  - Borsod-Abauj-Zemplen County Hospital and University Teaching Hospital, Miskolc, Borsod-Abauj Zemplen county
  - University of Pecs, Faculty of Medicine Neurosurgery Clinic, Pécs
  - University of Szeged, Faculty of Medicine, Pécs
- India (3):
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - CARE Hospital, Hyderabad
  - King Edward Memorial Hospital, Pune
- Israel (3):
  - Rambam Medical Centre, Haifa
  - Hadassah Universtity Medical Center, Jerusalem
  - Sheba Medical Centre, Tel Litwinsky
- Italy (4):
  - Osepedale Maggiore Bellaria, Bologna
  - Azienda Ospedaliera di Careggi, Florence
  - Azienda Osepedaliera San Giovanni - Addolorata, Rome
  - Ospedale Maggiore, Verona
- Mexico (2):
  - Instituto Nacional de Neurologia y Neurocirugia, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez" Universidad Autonoma de Nuevo Leon, Monterrey
- Elisabeth Ziekenhuis, Tilburg, Netherlands
- Norway (3):
  - Haukeland University Hospital, Helse Bergen HF, Bergen
  - Ulleval Univ Hosp, Oslo
  - Universitetssykehuset Nord-Norge, Tromsø
- Poland (2):
  - Szpital Akademii Medycznej w Gdansku, Gdansk
  - Samodzielny Publiczny Centralny Szpital Kliniczy w Warszawie, Warsaw
- Singapore (2):
  - National University Hospital, Singapore
  - National Neuroscience Institute, Singapore
- Slovenia (2):
  - University Clinical Centre Ljubljana, Ljubljana
  - General Hospital Maribor, Maribor
- Spain (5):
  - Hospital Vali d' Hebron, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Complejo Hospotalario Virgen de las Nieves-Hospital de Rehabilitacion y Traumatologia, Granada
  - Hospital Universitario 12 se Octubre, Madrid
  - Hospital de Son Dureta, Palma de Mallorca
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Linkoping University Hospital, Linköping
  - Lund University Hospital, Lund
- Switzerland (4):
  - Kantonsspital Aarau, Aarau
  - Universitatsklinik Bern, Bern
  - Geneva University Hospital, Geneva
  - Universitatsspital Zurich, Zurich
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Result] Macdonald RL, Higashida RT, Keller E, Mayer SA, Molyneux A, Raabe A, Vajkoczy P, Wanke I, Bach D, Frey A, Nowbakht P, Roux S, Kassell N. Randomized trial of clazosentan in patients with aneurysmal subarachnoid hemorrhage undergoing endovascular coiling. Stroke. 2012 Jun;43(6):1463-9. doi: 10.1161/STROKEAHA.111.648980. Epub 2012 Mar 8. PMID 22403047
- [Derived] Mayer SA, Aldrich EF, Bruder N, Hmissi A, Macdonald RL, Viarasilpa T, Marr A, Roux S, Higashida RT. Thick and Diffuse Subarachnoid Blood as a Treatment Effect Modifier of Clazosentan After Subarachnoid Hemorrhage. Stroke. 2019 Oct;50(10):2738-2744. doi: 10.1161/STROKEAHA.119.025682. Epub 2019 Aug 9. PMID 31394993